CLINICAL TRIAL: NCT07263282
Title: Left Atrium Strain as a Predictor of In-Hospital Outcomes in Patients With ST-Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: LA Strain in Predicting Early Complication in STEMI After PPCI
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Youssef Dandrawy, principle investigator, Assiut University
Other Study IDs: left atrial strain in STEMI
Record Dates: First submitted 2025-11-16; First posted 2025-12-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction
Keywords: strain in STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group normal strain: group normal parameters of LA strain by 2D echocardiography
  Interventions: Other: 2D echocardiography
- group low strain: group low parameters of LA strain by 2D echocardiography
  Interventions: Other: 2D echocardiography
- group control: control group to provide reference for normal parameters of LA strain for age by 2D echocardiography
  Interventions: Other: 2D echocardiography

INTERVENTIONS:
Other: 2D echocardiography — LA strain by 2D echocardiographic speckle tracking analysis

SUMMARY:
The goal of this observational study To evaluate the predictive value of left atrial strain for in-hospital outcomes in patients with ST-segment elevation myocardial infarction undergoing PPCI. The main questions it aims to answer are:

Is low parameters of left atrial strain associated early complication ? What is the correlation between LA strain parameters and conventional echocardiographic indices of left ventricular systolic and diastolic function ? Is there more affection to LA strain in certain territory over the others ? What is the correlation between LA strain and LA volume index across infarct territories ? Does LA strain Correlate with TAPSE and PASP to evaluate right-heart interactions ?

DETAILED DESCRIPTION:
The overall trend of ST-segment elevated myocardial infarction has shown an annual increase. Post-infarction heart failure is one of the major adverse cardiovascular events in patients with post-percutaneous coronary intervention.

Therefore, the prediction and accurate assessment of in-hospital outcomes in patients have gained more research and clinical attention.

Left ventricular ejection fraction may no longer be the sole and most reliable predictor of events after a STEMI. Left atrial function may be a comprehensive marker of left-sided cardiac function, as it reflects both diastolic and systolic properties of overall cardiac function.

LA function influences left ventricular filling and cardiac output. Compromised LV function leads to reduced passive LA stretch and filling, contributing to increased LV filling pressures and a subsequent decline in LA function and compliance.

. LA strain is a measurement of atrial myocardial deformation, which is less influenced by cardiac preload and less angle-dependent compared to volumetric indices, such as the left atrial volume index and E/e' ratio.

LA strain is useful in various clinical scenarios, as predicting atrial fibrillation, diastolic dysfunction, and as a measure of LV filling pressure .

LA strain by echocardiographic speckle tracking analysis, is relatively inexpensive, non-invasive and easy to perform, so may be useful as a predictor of in-hospital outcomes.

Previous studies have demonstrated that reduced LA function is linked to clinical outcomes including all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Diagnosed with ST-segment elevation myocardial infarction (STEMI) according to current ESC/AHA criteria
* Underwent successful primary percutaneous coronary intervention (PPCI) within 12 hours of symptom onset.
* Sinus rhythm on admission .
* Trans thoracic echocardiography (TTE) performed within 48 hours of admission with adequate image quality for speckle-tracking analysis.

Exclusion Criteria:

* Previous myocardial infarction or prior PCI/CABG.
* Patients known to have atrial fibrillation or other sustained supraventricular arrhythmias.
* Significant valvular heart disease (severe stenosis or regurgitation).
* Congenital heart disease or cardiomyopathy (hypertrophic, dilated, restrictive).
* Poor echocardiographic window preventing LA strain analysis .
* Mechanical complications (e.g., papillary muscle rupture, VSD, free wall rupture).
* Prior cardiac surgery or known structural lesions that preventing reliable LA measurement.
* patient presenting with killip class III or IV from the start

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with ST-segment elevation myocardial infarction and Underwent successful primary percutaneous coronary intervention and control group to provide baseline parameters for comparing LA strain and other echocardiographic parameters
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
the predictive value of left atrial strain for detecting incidence of in-hospital outcomes in patients with ST-segment elevation myocardial infarction undergoing primary PCI. | up to one week
  To evaluate the predictive value of left atrial strain for hospitalized patients with ST-segment elevation myocardial infarction undergoing primary PCI as regarding
  * All-cause in-hospital mortality
  * New/worsening heart failure requiring IV therapy or ICU care
  * Cardiogenic shock (requiring inotropes or mechanical support)
  * Sustained ventricular arrhythmia (VT/VF)

SECONDARY OUTCOMES:
correlation with other parameters | up to one week
  Correlation between LA strain parameters (reservoir, conduit, and contractile strain) by speckle tracking echocardiography and conventional echocardiographic indices of left ventricular (LV) systolic and diastolic function (LVEF, LVGLS , E/e', LAVI).
LA strain across different territories | up to one week
  Compare LA strain (reservoir, conduit, contractile) by speckle tracking echocardiography between anterior (LAD-territory) vs inferior (RCA/LCx-territory) STEMI as which territory would have more affection to LA strain
LA stain vs LAVI | up to one week
  Correlation between LA strain and LA volume index (LAVI) across infarct territories
LA strain and right side | up to one week
  Correlate LA strain with TAPSE and PASP to evaluate right-heart interactions

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Fouad, Professor, Principal Investigator — Assiut University; Magdy I Algowhary, Assistant Professor, Principal Investigator — Assiut University; Ahmed G Bakry, Assistant Professor, Principal Investigator — South Valley University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Badano LP, Kolias TJ, Muraru D, Abraham TP, Aurigemma G, Edvardsen T, D'Hooge J, Donal E, Fraser AG, Marwick T, Mertens L, Popescu BA, Sengupta PP, Lancellotti P, Thomas JD, Voigt JU; Industry representatives; Reviewers: This document was reviewed by members of the 2016-2018 EACVI Scientific Documents Committee. Standardization of left atrial, right ventricular, and right atrial deformation imaging using two-dimensional speckle tracking echocardiography: a consensus document of the EACVI/ASE/Industry Task Force to standardize deformation imaging. Eur Heart J Cardiovasc Imaging. 2018 Jun 1;19(6):591-600. doi: 10.1093/ehjci/jey042. PMID 29596561
- [Result] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982
- [Result] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Result] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Result] Ahmeti A, Bytyci FS, Bielecka-Dabrowa A, Bytyci I, Henein MY. Prognostic value of left atrial volume index in acute coronary syndrome: A systematic review and meta-analysis. Clin Physiol Funct Imaging. 2021 Mar;41(2):128-135. doi: 10.1111/cpf.12689. Epub 2021 Jan 12. PMID 33372377
- [Result] Wu H, Wang H, Wang X, Xu L, Wu J. Myocardial strain combined with clinical risk factors in the prediction of in-hospital heart failure among patients with ST-segment elevation myocardial infarction. Clin Radiol. 2024 Nov;79(11):e1304-e1311. doi: 10.1016/j.crad.2024.07.016. Epub 2024 Jul 26. PMID 39191561
- [Result] Chu AA, Wu TT, Zhang L, Zhang Z. The prognostic value of left atrial and left ventricular strain in patients after ST-segment elevation myocardial infarction treated with primary percutaneous coronary intervention. Cardiol J. 2021;28(5):678-689. doi: 10.5603/CJ.a2020.0010. Epub 2020 Feb 10. PMID 32037499
- [Result] Svartstein AW, Lassen MH, Skaarup KG, Grove GL, Vyff F, Ravnkilde K, Pedersen S, Galatius S, Modin D, Biering-Sorensen T. Predictive value of left atrial strain in relation to atrial fibrillation following acute myocardial infarction. Int J Cardiol. 2022 Oct 1;364:52-59. doi: 10.1016/j.ijcard.2022.05.026. Epub 2022 May 14. PMID 35577164
- [Result] Nagueh SF, Khan SU. Left Atrial Strain for Assessment of Left Ventricular Diastolic Function: Focus on Populations With Normal LVEF. JACC Cardiovasc Imaging. 2023 May;16(5):691-707. doi: 10.1016/j.jcmg.2022.10.011. Epub 2023 Jan 11. PMID 36752445
- [Result] Robinson S, Ring L, Oxborough D, Harkness A, Bennett S, Rana B, Sutaria N, Lo Giudice F, Shun-Shin M, Paton M, Duncan R, Willis J, Colebourn C, Bassindale G, Gatenby K, Belham M, Cole G, Augustine D, Smiseth OA. The assessment of left ventricular diastolic function: guidance and recommendations from the British Society of Echocardiography. Echo Res Pract. 2024 Jun 3;11(1):16. doi: 10.1186/s44156-024-00051-2. PMID 38825710
- [Result] Li R, Sun F, Piao S, He X, Li R, Xu L, Song G, Cong J. Left Atrial Strain and Compliance Correlate with Diastolic Dysfunction Grades and Complications during Pre-eclampsia: A Speckle-Tracking Echocardiography Study. Ultrasound Med Biol. 2021 Dec;47(12):3411-3419. doi: 10.1016/j.ultrasmedbio.2021.08.003. Epub 2021 Aug 27. PMID 34456083
- [Result] Lenselink C, Ricken KWLM, Groot HE, de Bruijne TJ, Hendriks T, van der Harst P, Voors AA, Lipsic E. Incidence and predictors of heart failure with reduced and preserved ejection fraction after ST-elevation myocardial infarction in the contemporary era of early percutaneous coronary intervention. Eur J Heart Fail. 2024 May;26(5):1142-1149. doi: 10.1002/ejhf.3225. Epub 2024 Apr 4. PMID 38576163
- [Result] Zhang L, Liu Z, Zhu Y, Wu M, Huang H, Yang W, Peng K, Zeng J. Development and validation of a prognostic model for predicting post-discharge mortality risk in patients with ST-segment elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PPCI). J Cardiothorac Surg. 2024 Mar 30;19(1):163. doi: 10.1186/s13019-024-02665-3. PMID 38555468
- [Result] Abe T, Olanipekun T, Adedinsewo D, Ogunmoroti O, Udongwo N, Effoe V, Rice B, Onuorah I, Ghali JK, Mehta PK, Michos ED. Trends and Outcomes of ST-Segment-Elevation Myocardial Infarction Among Young Women in the United States. J Am Heart Assoc. 2023 Mar 7;12(5):e026811. doi: 10.1161/JAHA.122.026811. Epub 2023 Feb 27. PMID 36847058